CLINICAL TRIAL: NCT01888822
Title: Ciprofloxacin, Ampicillin-sulbactam and Placebo Prophylaxis in Laparoscopic Cholecystectomy. A Randomized Controlled Study
Brief Title: Antibiotic Prophylaxis in Laparoscopic Cholecystectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Erasmo Spaziani, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MarPic63
Record Dates: First submitted 2013-06-13; First posted 2013-06-28 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cholelithiasis
Keywords: Laparoscopic cholecystectomy; Prophylactic antibiotics
MeSH Terms: conditions — Cholelithiasis | interventions — Ciprofloxacin; sultamicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Intravenous infusion of 0.9% Sodium Chloride 250 ml during induction of anesthesia and before laparoscopic cholecystectomy.
  Interventions: Drug: Placebo
- Ampicillin-sulbactam (Active Comparator): Intravenous infusion of 3gr ampicillin-sulbactam in 0.9% Sodium Chloride 250 ml during induction of anesthesia and before laparoscopic cholecystectomy.
  Interventions: Drug: Ampicillin-sulbactam
- Ciprofloxacin (Active Comparator): Intravenous infusion of 400 mg ciprofloxacin in 0.9% Sodium Chloride 250 ml during induction of anesthesia and before laparoscopic cholecystectomy.
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin — Prophylactic ciprofloxacin infusion before elective laparoscopic cholecystectomy
  Arms: Ciprofloxacin
Drug: Ampicillin-sulbactam — Prophylactic ampicillin-sulbactam infusion before elective laparoscopic cholecystectomy
  Arms: Ampicillin-sulbactam
Drug: Placebo — Prophylactic placebo infusion before elective laparoscopic cholecystectomy
  Arms: Placebo

SUMMARY:
The trial aims to assess the value of two-regimen antibiotic prophylaxis versus placebo in elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
All patients enrolled will be submitted to laparoscopic cholecystectomy. The primary aim of the trial will be to assess the role of prophylactic i.v. infusion of ampicillin-sulbactam, ciprofloxacin, and placebo to reduce the rate of surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic cholecystectomy;
* patients suffering from gallbladder stones,chronic cholecystitis, cholesterolosis, or gallbladder polyps.

Exclusion Criteria:

* acute cholecystitis;
* acute cholangitis;
* acute pancreatitis;
* pregnant or lactating women;
* antibiotic allergy;
* antibiotic therapy within 48 hours to 7 days prior to surgery;
* clinically active infection at the moment of surgery;
* evidence of common bile duct stones;
* contraindications for laparoscopic cholecystectomy;
* no other additional procedure;
* indication of obligatory antibiotic prophylaxis because the medical condition was different from biliary disease (immunosuppression, corticoid use, etc).
* patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days after operation
  Surgical site infection defined according to the Centre of Disease Control (CDC) classification, recorded as 'yes' or 'no'.

SECONDARY OUTCOMES:
Extra-abdominal infections | 30 days
  Extra-abdominal infections defined according to the CDC classification, recorded as 'yes' or 'no'.
Adverse events. | 30 days
  Adverse events, defined as allergic reactions to antibiotics.
Quality of life | 30 days
  Quality of life measured with the 36-Item Short Form Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Erasmo Spaziani, MD, PhD, Study Director — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome- Polo Pontino, Terracina, Latina, Italy

REFERENCES:
- [Background] Sanabria A, Dominguez LC, Valdivieso E, Gomez G. Antibiotic prophylaxis for patients undergoing elective laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2010 Dec 8;2010(12):CD005265. doi: 10.1002/14651858.CD005265.pub2. PMID 21154360